CLINICAL TRIAL: NCT04377919
Title: Effects of Cranberry Supplementation on Chronic Kidney Disease Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DeniseMafra6
Record Dates: First submitted 2018-09-28; First posted 2020-05-07 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Renal Insufficiency, Chronic; Inflammation; Oxidative Stress; Gastrointestinal Microbiome
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry (Active Comparator): Administration of 2 capsules with 500mg (Miralys Ltda) of cranberry extract per day, for 8 weeks
  Interventions: Dietary Supplement: Cranberry
- Placebo (Placebo Comparator): Administration of 2 capsules with 500mg of maize starch per day, for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cranberry — The patients will receive 2 capsules per day containing 500mg of cranberry extract for 8 weeks
  Arms: Cranberry
Dietary Supplement: Placebo — The patients will receive 2 capsules per day containing 500mg of maize starch for 8 weeks
  Arms: Placebo

SUMMARY:
Patients with chronic kidney disease (CKD) have several complications that are linked to oxidative stress and inflammation, and among the most recently studied is the alteration of the intestinal microbiota. Considering this scenario, bioactive compounds have been considered as a therapeutic alternative in the modulation of intestinal microbiota as well as transcription factors such as nuclear-kappa factor B (NF-κB) and factor 2 nuclear factor-related erythroid 2 Nrf2), involved with oxidative stress and inflammation. Among several foods, cranberry is a fruit rich in flavonoids and other polyphenols, which has antioxidant, anti-inflammatory and immunoregulatory actions and may be an adjuvant treatment for CKD complications. However, clinical evidence evaluating the effects of cranberry is limited and there are no studies specifically involving patients with CKD. Thus, the present randomized crossover double-blind crossover with placebo-controlled washout period will aim to evaluate the effects of cranberry supplementation on the modulation of the intestinal microbiota and expression of transcription factors as well as cytokine levels inflammatory effects of CKD patients.

DETAILED DESCRIPTION:
This is a longitudinal study with a randomized crossover design, double-blind, placebo-controlled, and with washout period. Thirty non-dialysis patients of both genders, aged between 18 and 60 years and with CKD stage3-4 (glomerular filtration rate < 59 mL/min/1.73 m2) will be included in the study. Pregnant patients, smokers and those under use of antibiotics in the last 3 months, or in use antithrombotic, pre-, pro- or synbiotic supplements, antioxidant supplements or habitual cranberry intake will be excluded. In addition, those with autoimmune and infectious diseases, cancer, liver diseases and HIV will also not be included in the study. The patients that fulfill the eligible criteria and sign the ethical informed consent will be randomized to either Group A (Cranberry) or Group B (Placebo). During 12 weeks, patients allocated in group A will receive capsules containing cranberry extract (Vaccinium macrocarpon to 25% anthocyanosides 160mg, equivalent to 40mg anthocyanosides), once daily (lunch), totaling 500mg / day and those allocated in the group B will receive a placebo (500mg of corn starch). After the supplementation period, a 12-week washout will be performed for subsequent crossover of the supplement. The randomization will be computed in the ratio of 1: 1, with block size of 15 (Cranberry group and Control), to receive cranberry or placebo. This project was approved by the Ethics Committee of the Faculty of Medicine-UFF, n. 2.653.752.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Kidney Disease in conservative treatment
* Aged 18 years or older
* Must be able to swallow tablets

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last 3 months
* Using antioxidant supplements in the last 3 months
* Usual intake of cranberry fruit or extract
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Antioxidants and anti-inflammatory biomarkers | 3 months
  Evaluate the supplementation effects in anti-inflammatory biomarkers- Nrf2 and antioxidants enzymes
Inflammatory biomarkers | 3 months
  Evaluate the supplementation effects in inflammatory biomarkers- factor nuclear kappa B (NFkB), interleukin 6 (IL-6), tumor necrosis factor alpha (TNF-alpha)
Biochemical Routine | 12 weeks
  Urea, creatinine, albumin, lipid profile plasma levels
Uremic toxins | 6 months
  P-cresol, indoxyl sulfate plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, phd, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Souza Gouveia Moreira L, Resende Teixeira KT, Cardozo LFMF, Alvarenga L, Regis B, Sousa de Brito J, de Oliveira Leal V, Borges NA, de Souza da Costa Brum I, Carraro-Eduardo JC, Borini GB, Berretta AA, Ribeiro-Alves M, Mafra D. Effects of Cranberry Extract (Vaccinium macrocarpon) Supplementation on Lipid Peroxidation and Inflammation in Patients with Chronic Kidney Disease (Stages 3-4): A Randomized Controlled Trial. J Nutr Metab. 2024 May 8;2024:9590066. doi: 10.1155/2024/9590066. eCollection 2024. PMID 38752013